CLINICAL TRIAL: NCT01063374
Title: Low Glycemic Index Diets to Improve Glycemic Control and Cardiovascular Disease in Type 2 Diabetics
Brief Title: Low Glycemic Index Diet for Type 2 Diabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, David Jenkins, Principle Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-193
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low glycemic index, diabetic diet (Active Comparator): low glycemic index, diabetic diet
  Interventions: Dietary Supplement: low glycemic diet instruction
- high cereal fibre, diabetic diet (Active Comparator): high cereal fibre, diabetic diet
  Interventions: Dietary Supplement: high cereal fibre diet instruction

INTERVENTIONS:
Dietary Supplement: low glycemic diet instruction
  Arms: low glycemic index, diabetic diet
Dietary Supplement: high cereal fibre diet instruction
  Arms: high cereal fibre, diabetic diet

SUMMARY:
A low glycemic index diet may improve glycemic control and reduce plaque buildup in arteries of those with type 2 diabetes. Subjects will be randomly assigned to receive dietary advice on either a low glycemic index diet, or a high cereal fibre diet, for three years.

DETAILED DESCRIPTION:
All subjects will be randomized to one 3-year treatment in a two-treatment parallel design.

Treatments:

1. low glycemic index dietary advice (e.g. to eat intact grain cereals, parboiled rice, cracked wheat, pasta, peas, beans, lentils, and baked goods made from legume flour); or
2. a high cereal fiber diet emphasizing whole grains. Duration: The study will consist of approximately two months of recruitment and patient selection, during which time estimation of individual caloric requirements will be assessed, and a 3 year treatment period assigned.

Study Details: Fasting blood samples are obtained at screening, week -2, and months 0, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36 each study period. HbA1c will be assessed on all visits. A carotid ultrasound (CUS) (screening, months 0, 12 and 36) and magnetic resonance imaging (MRI) (months 0, 12 and 36) technologies will be used to assess arterial wall thickening and changes in the nature of carotid plaques. Twenty-four hour urine for urinary C-peptide analyses will be obtained immediately prior to the beginning of the study and at the end of each 3 year treatment phase. At the end of the 3 year treatment period, subjects who wish to undertake the alternate treatment will be given appropriate instruction.

ELIGIBILITY:
Inclusion Criteria:

Men and women with type 2 diabetes who

* are treated with oral hypoglycemic agents at a stable dose for at least 8 weeks
* have a HbA1c in the range of 6.5 to 8.0% at screening and at the prestudy visit
* have diabetes diagnosed >6 months
* have maintained stable weight for 2 months (within 3%)
* have a valid OHIP card and a family physician
* if prescribed lipid medication, have taken a stable dose for at least 2 weeks
* if prescribed blood pressure medication, have taken a stable dose for at least 1 week
* can keep written food records, with the use of a digital scale

Exclusion Criteria: Individuals who

* take insulin
* take steroids
* have GI disease (gastroparesis, celiac disease, ulcerative colitis, Crohn's Disease, IBS)
* have had a major cardiovascular event (stroke or myocardial infarction) in the past 6 months
* take warfarin (Coumadin)
* have had major surgery in the past 6 months
* have a major debilitating disorder
* have clinically significant liver disease (AST or ALT > 130 U/L), excluding NAFL or NASH
* have hepatitis B or C
* have renal failure (high creatinine > 150 mmol/L)
* have serum triglycerides ≥ 6.0 mmol/L
* have a history of cancer, except non-melanoma skin cancer (basal cell, squamous cell)
* have food allergies to study food components
* have elevated blood pressure (> 145/90) unless approved by GP
* have acute or chronic infections (bacterial or viral)
* have chronic inflammatory diseases (e.g. rheumatoid arthritis, lupus; ulcerative colitis)
* have other conditions which in the opinion of any of the investigators would make them unsuitable for the study
* If HbA1c rises above 8.5% over two consecutive routine measurements, subjects will be referred back to their family doctors for an increase in anti hyperglycemic medications according to a predetermined protocol.
* Any condition or circumstance which would prevent an individual from having an MRI (e.g. individuals with prostheses or metal implants, or those who are excessively claustrophobic)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-03; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
plaque volume | 1, 3 years

SECONDARY OUTCOMES:
intima media thickness | 0, 1, and 3 years
plaque morphology | 0, 1, 3 years
HbA1c | every 3 months for 3 years
serum lipids | every 3 months for 3 years
blood pressure | every 3 months for 3 years
serum fasting glucose | creatinine, urea, and C-peptides in 24 hour urine collection
anthropometric measures (weight, waist and hip circumference) | every 3 months for 3 years
retinal photography | 1, 3 years
  ophthalmological assessment using fundoscopy

CONTACTS AND LOCATIONS:
Overall Officials: David Mazer, Study Chair — St. Michael's Hospital Research Ethics Board
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Clinical Nutrition & Risk Factor Modification Centre, St. Michael's Hospital Health Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiavaroli L, Mirrahimi A, Ireland C, Mitchell S, Sahye-Pudaruth S, Coveney J, Olowoyeye O, Patel D, de Souza RJ, Augustin LS, Bashyam B, Pichika SC, Blanco Mejia S, Nishi SK, Leiter LA, Josse RG, McKeown-Eyssen GE, Moody AR, Kendall CW, Sievenpiper JL, Jenkins DJ. Cross-sectional associations between dietary intake and carotid intima media thickness in type 2 diabetes: baseline data from a randomised trial. BMJ Open. 2017 Mar 22;7(3):e015026. doi: 10.1136/bmjopen-2016-015026. PMID 28336747
- [Derived] Chiavaroli L, Mirrahimi A, Ireland C, Mitchell S, Sahye-Pudaruth S, Coveney J, Olowoyeye O, Maraj T, Patel D, de Souza RJ, Augustin LS, Bashyam B, Blanco Mejia S, Nishi SK, Leiter LA, Josse RG, McKeown-Eyssen G, Moody AR, Berger AR, Kendall CW, Sievenpiper JL, Jenkins DJ. Low-glycaemic index diet to improve glycaemic control and cardiovascular disease in type 2 diabetes: design and methods for a randomised, controlled, clinical trial. BMJ Open. 2016 Jul 7;6(7):e012220. doi: 10.1136/bmjopen-2016-012220. PMID 27388364